CLINICAL TRIAL: NCT01390584
Title: Phase II Trial of Response-Adapted Therapy Based on Positron Emission Tomography (PET) for Bulky Stage I and II Classical Hodgkin Lymphoma (HL)
Brief Title: Chemotherapy Based on PET Scan in Treating Patients With Stage I or Stage II Hodgkin Lymphoma
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: slow accrual
Sponsor: ECOG-ACRIN Cancer Research Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Organization: Eastern Cooperative Oncology Group (Network)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: E2410; NCT01390584 (Registry Identifier: ClinicalTrials.gov); U01CA079778 (NIH); U01CA080098 (NIH)
Record Dates: First submitted 2011-07-07; First posted 2011-07-11 (Estimated); Results first posted 2020-12-22 (Actual); Last update posted 2023-06-29 (Actual); Status verified 2023-06

CONDITIONS: Lymphoma
Keywords: stage I adult Hodgkin lymphoma; stage II adult Hodgkin lymphoma
MeSH Terms: conditions — Lymphoma; Hodgkin Disease | interventions — Doxorubicin; Bleomycin; Vinblastine; Positron Emission Tomography Computed Tomography; Dacarbazine; Etoposide; Podophyllotoxin; Cyclophosphamide; Vincristine; Procarbazine; Prednisone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- ABVD + INRT (Experimental): Induction ABVD chemotherapy: Patients receive doxorubicin hydrochloride IV, bleomycin sulfate IV, vinblastine IV over 3-5 minutes, and dacarbazine IV over 30 minutes on days 1 and 15. Treatment repeats every 28 days for 2 courses.
  PET-CT scan: Then patients undergo fludeoxyglucose F 18 (18 FDG) positron emission tomography (PET)/computed tomography (CT). If results are negative, patients receive the following treatment.
  ABVD + INRT: Patients receive doxorubicin hydrochloride, bleomycin sulfate, vinblastine, and dacarbazine as in induction chemotherapy. Treatment repeats every 28 days for 4 courses. Within 3-6 weeks after completion of chemotherapy, patients undergo involved-node radiotherapy (INRT) 5 days a week for approximately 3½ weeks.
  Interventions: Drug: Doxorubicin; Drug: Bleomycin; Drug: Vinblastine; Diagnostic Test: PET; Radiation: INRT; Drug: Dacarbazine
- ABVD + BEACOPP + INRT (Experimental): Induction ABVD chemotherapy: Patients receive doxorubicin hydrochloride IV, bleomycin sulfate IV, vinblastine IV over 3-5 minutes, and dacarbazine IV over 30 minutes on days 1 and 15. Treatment repeats every 28 days for 2 courses.
  PET-CT scan: Then patients undergo fludeoxyglucose F 18 (18 FDG) positron emission tomography (PET)/computed tomography (CT). If results are positive, patients receive the following treatment.
  BEACOPP + INRT: Patients receive doxorubicin hydrochloride IV and cyclophosphamide IV over 60 minutes on day 1, etoposide IV over 60 minutes on days 1-3, procarbazine hydrochloride orally (PO) on days 1-7, prednisone PO on days 1-14, and bleomycin sulfate IV and vincristine sulfate IV on day 8. Treatment repeats every 21 days for 4 courses. Within 3-6 weeks after completion of chemotherapy, patients who achieve complete response with a negative 18FDG-PET/CT scan undergo INRT 5 days a week for approximately 3½ weeks.
  Interventions: Drug: Doxorubicin; Drug: Bleomycin; Drug: Vinblastine; Diagnostic Test: PET; Radiation: INRT; Drug: Dacarbazine; Drug: Etoposide; Drug: Cyclophosphamide; Drug: Vincristine; Drug: Procarbazine; Drug: Prednisone

INTERVENTIONS:
Drug: Doxorubicin — IV
  Other Names: Adriamycin R; Rubex R; Adriamycin RDF R; Adriamycin PFS R; hydroxydaunorubicin; hydroxydaunomycin; ADR
Drug: Bleomycin — IV
  Other Names: Blenoxane R; BLM; Bleo
Drug: Vinblastine — IV
  Other Names: Velban R; vinblastine sulfate; vincaleukoblastine; VLB; Velsar R; Alkaban AQ R
Diagnostic Test: PET — fludeoxyglucose F 18 Imaging exam
  Other Names: PET/CT
Radiation: INRT — selective external radiation therapy
Drug: Dacarbazine — IV
  Other Names: DTIC; DTIC-Dome®; DIC; imidazole carboxamide; dimethyl triazeno imidazole carboxamide; NSC # 45388
Drug: Etoposide — IV
  Other Names: VP-16; VePesidÒ; VP-16-213; EPEG; epipodophyllotoxin; NSC #141540
  Arms: ABVD + BEACOPP + INRT
Drug: Cyclophosphamide — May be given orally, IV push, or by IV infusion
  Other Names: CytoxanÒ; NeosarÒ; CTX; CPM
  Arms: ABVD + BEACOPP + INRT
Drug: Vincristine — IV
  Other Names: Oncovin R; Vincasar PFS R; vincristine sulfate; VCR; leucocristine; LCR
  Arms: ABVD + BEACOPP + INRT
Drug: Procarbazine — PO
  Other Names: MatulaneR; Ibenzmethyzin; Natulanar; N-Methylhydrazine
  Arms: ABVD + BEACOPP + INRT
Drug: Prednisone — PO
  Other Names: Deltasone; Orasone; Medicorten; Panasol-S; Liquid-Pred
  Arms: ABVD + BEACOPP + INRT

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as doxorubicin hydrochloride, bleomycin sulfate, vinblastine, dacarbazine, cyclophosphamide, etoposide, procarbazine hydrochloride, vincristine sulfate, and prednisone, work in different ways to stop the growth of cancer cells, either by killing the cells or by stopping them from dividing. Radiation therapy uses high-energy x rays to kill cancer cells. Giving combination chemotherapy together with radiation therapy may kill more cancer cells. Comparing results of imaging procedures, such as PET scans and CT scans, done before, during, and after chemotherapy may help doctors predict a patient's response to treatment and help plan the best treatment.

PURPOSE: This phase II clinical trial studies how well chemotherapy based on PET/CT scan works in treating patients with stage I or stage II Hodgkin lymphoma.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* To evaluate the progression-free survival (PFS) at 36 months following registration for patients who are positron emission tomography (PET) negative after 2 courses of ABVD, and receive 4 additional courses of doxorubicin hydrochloride, bleomycin sulfate, vinblastine, and dacarbazine (ABVD) followed by involved-nodal radiotherapy [INRT] of 30-30.6 Gy.

Secondary

* To evaluate the PET-negative rate after 2 courses of ABVD chemotherapy in patients with stage I/II Hodgkin lymphoma with bulky mediastinal disease.
* To evaluate the PFS at 36 months for patients who are PET positive after 2 courses of chemotherapy and receive 4 courses of escalated bleomycin sulfate, etoposide, doxorubicin hydrochloride, cyclophosphamide, vincristine sulfate, procarbazine hydrochloride, and prednisone (BEACOPP) followed by INRT of 30-30.6 Gy.
* To evaluate the complete response (CR) rate and overall survival (OS) for PET-positive and PET-negative patients after 2 courses of ABVD.
* To identify sites of relapse following combined-modality therapy (CMT) for patients with large mediastinal adenopathy and correlate with RT fields.
* To assess toxicity on both arms of study.
* To assess reproductive function at baseline and at 3 years after ABVD or escalated BEACOPP with specific serum markers.
* To bank serum and plasma at baseline and selected time points to assess the prognostic value of various markers such as, but not limited to, SCD30, IL10, CCL17, CCL22, and MDC.
* To create tissue microarrays (TMAs) from patient tumor blocks for future biomarker assessment including, but not limited to, bcl-2, FOXP3, and macrophage content.
* To measure serum TARC levels pre-treatment and post two courses of ABVD and correlate with PET-CT findings (performed at same time points) and 3 year PFS.

Tertiary

* To assess the predictive value of fludeoxyglucose F 18 (18FDG) uptake, as measured by semi-quantitative measurements including standard uptake variables (SUVs), with respect to response at the end of chemotherapy and PFS.
* To compare the predictive value for response and PFS of FDG uptake alone to that of FDG uptake in combination with CT size change information.
* To compare the predictive value for response and PFS of FDG uptake alone to that of FDG uptake in combination with available serum and tissue molecular biomarkers.
* To compare the results of the secondary imaging objectives with the corresponding CALGB 50801 results (contingent on reaching agreement with CALGB on the combined analysis of the two studies).

OUTLINE: This is a multicenter study.

Induction ABVD chemotherapy: Patients receive doxorubicin hydrochloride IV, bleomycin sulfate IV, vinblastine IV over 3-5 minutes, and dacarbazine IV over 30 minutes on days 1 and 15. Treatment repeats every 28 days for 2 courses in the absence of disease progression or unacceptable toxicity.

Patients are then assigned to an intervention arm according to fludeoxyglucose F 18 (18 FDG) positron emission tomography (PET)/computed tomography (CT) results (negative vs positive).

* ABVD (18FDG-PET/CT negative): Patients receive doxorubicin hydrochloride, bleomycin sulfate, vinblastine, and dacarbazine as in induction chemotherapy. Treatment repeats every 28 days for 4 courses in the absence of disease progression or unacceptable toxicity. Within 3-6 weeks after completion of chemotherapy, patients undergo involved-node radiotherapy (INRT) 5 days a week for approximately 3½ weeks.
* Escalated or standard BEACOPP* (18FDG-PET/CT positive): Patients receive doxorubicin hydrochloride IV and cyclophosphamide IV over 60 minutes on day 1, etoposide IV over 60 minutes on days 1-3, procarbazine hydrochloride orally (PO) on days 1-7, prednisone PO on days 1-14, and bleomycin sulfate IV and vincristine sulfate IV on day 8. Treatment repeats every 21 days for 4 courses in the absence of disease progression or unacceptable toxicity. Within 3-6 weeks after completion of chemotherapy, patients who achieve complete response with a negative 18FDG-PET/CT scan undergo INRT 5 days a week for approximately 3½ weeks.

NOTE: *HIV-positive patients whose 18FDG-PET/CT scans are positive after two courses of induction ABVD receive 4 courses of standard BEACOPP followed by INRT.

Patients undergo 18FDG-PET scans at baseline, and within 8-10 days after 2 courses of ABVD induction chemotherapy. Patients also undergo 18FDG-PET/CT** scan within 3-8 weeks after completion of 4 courses of BEACOPP and 6 courses of ABVD, and 3 months after completion of INRT.

NOTE: **If PET/CT remains positive, then a biopsy may be performed if medically appropriate or clinically feasible at the discretion of the treating physician. If biopsy is positive, patients will be followed for survival and secondary malignancies or new primaries.

Patients may undergo blood sample collection for correlative studies.

After completion of study therapy, patients are followed up every 3 months for 1 year, every 6 months for 2 years, and then annually for up to 10 years.

ELIGIBILITY:
Inclusion Criteria:

* Histologically proven classical Hodgkin lymphoma subclassified according to the World Health Organization (WHO) Classification of Tumors, 4th edition (2008)
* Patients must have clinical stage IA, IB, IIA, or IIB disease

  * Patients with "E" extensions will be eligible if all other criteria have been met
* Patients must have a mediastinal mass > 0.33-cm maximum intrathoracic diameter on standing postero-anterior chest x-ray or measuring > 10 cm in its largest diameter on axial CT images
* Bone marrow biopsy is required
* ECOG performance status 0-2
* ANC ≥ 1,000/μL
* Platelet count ≥ 100,000/μL
* Hemoglobin ≥ 10 g/dL
* Serum creatinine ≤ 2 mg/dL
* Direct bilirubin ≤ 2 mg/dL
* AST/ALT ≤ 2 times upper limit of normal
* Women of childbearing potential and sexually active males must be strongly advised to use an accepted and effective method of contraception
* LVEF by ECHO or MUGA normal unless thought to be disease related
* DLCO ≥ 60% with no symptomatic pulmonary disease unless thought to be disease related
* Patients with a history of intravenous drug abuse, or any behavior associated with an increased risk of HIV infection, should be tested for exposure to the HIV virus, and an HIV test is required for entry on this protocol
* HIV-positive patients are eligible if they have CD4 counts ≥ 400/mm³ and are on concurrent antiretrovirals

  * Patient HIV status must be known prior to registration
  * HIV-positive patients must not have multi-drug resistant HIV infections; CD4 counts < 400/mm³; or other concurrent AIDS-defining conditions
* Concurrent antiretroviral therapy for HIV-positive patients (CD4 counts ≥ 400/mm³) allowed

Exclusion Criteria:

* Nodular lymphocyte-predominant Hodgkin lymphoma
* Pregnant or nursing
* "Currently active" second malignancy other than non-melanoma skin cancers

  * Patients are not considered to have a "currently active" malignancy if they have completed therapy and are considered by their physician to be at less than 30% risk of relapse
* Prior treatment (chemotherapy or radiation therapy) for Hodgkin lymphoma

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2013-05-24 (Actual); Primary Completion 2015-04-09 (Actual); Study Completion 2018-05-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ranjana Advani, MD, Study Chair — Stanford University
Locations (2):
- United States (2):
  - Stanford Cancer Center, Stanford, California
  - McGlinn Family Regional Cancer Center at Reading Hospital and Medical Center, Reading, Pennsylvania

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data may be made available upon request as per the ECOG-ACRIN Data Sharing Policy.

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was activated on April 2, 2012, accrued its first patient on May 24, 2013, and closed on January 24, 2014 with a final accrual of 6 patients.
Groups:
- Induction ABVD: Induction ABVD chemotherapy: Patients receive doxorubicin hydrochloride IV, bleomycin sulfate IV, vinblastine IV over 3-5 minutes, and dacarbazine IV over 30 minutes on days 1 and 15. Treatment repeats every 28 days for 2 courses.
Period: Step 1: Induction Tx (ABVD Then PET/CT)
Arm/Group | ABVD + INRT | ABVD + BEACOPP + INRT | Induction ABVD
Started | 4 | 1 | 1
Completed | 4 | 1 | 0
Not Completed | 0 | 0 | 1
Not completed — Ineligible | 0 | 0 | 1
Period: Step 2: ABVD or BEACOPP Then INRT
Arm/Group | ABVD + INRT | ABVD + BEACOPP + INRT | Induction ABVD
Started | 4 | 1 | 0
Completed | 4 | 1 | 0
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Only eligible and treated patients are included.
Groups:
- Arm A (ABVD + INRT): Induction ABVD chemotherapy: Patients receive doxorubicin hydrochloride IV, bleomycin sulfate IV, vinblastine IV over 3-5 minutes, and dacarbazine IV over 30 minutes on days 1 and 15. Treatment repeats every 28 days for 2 courses.
  PET-CT scan: Then patients undergo fludeoxyglucose F 18 (18 FDG) positron emission tomography (PET)/computed tomography (CT). If results are negative, patients receive the following treatment.
  ABVD + INRT: Patients receive doxorubicin hydrochloride, bleomycin sulfate, vinblastine, and dacarbazine as in induction chemotherapy. Treatment repeats every 28 days for 4 courses. Within 3-6 weeks after completion of chemotherapy, patients undergo involved-node radiotherapy (INRT) 5 days a week for approximately 3½ weeks.
- Arm B (ABVD + BEACOPP + INRT): Induction ABVD chemotherapy: Patients receive doxorubicin hydrochloride IV, bleomycin sulfate IV, vinblastine IV over 3-5 minutes, and dacarbazine IV over 30 minutes on days 1 and 15. Treatment repeats every 28 days for 2 courses.
  PET-CT scan: Then patients undergo fludeoxyglucose F 18 (18 FDG) positron emission tomography (PET)/computed tomography (CT). If results are positive, patients receive the following treatment.
  BEACOPP + INRT: Patients receive doxorubicin hydrochloride IV and cyclophosphamide IV over 60 minutes on day 1, etoposide IV over 60 minutes on days 1-3, procarbazine hydrochloride orally (PO) on days 1-7, prednisone PO on days 1-14, and bleomycin sulfate IV and vincristine sulfate IV on day 8. Treatment repeats every 21 days for 4 courses. Within 3-6 weeks after completion of chemotherapy, patients who achieve complete response with a negative 18FDG-PET/CT scan undergo INRT 5 days a week for approximately 3½ weeks.
- Total: Total of all reporting groups
Arm/Group | Arm A (ABVD + INRT) | Arm B (ABVD + BEACOPP + INRT) | Total
Number analyzed (Participants) | 4 | 1 | 5
Age, Continuous [Median (Full Range); unit: years] | 40 [39 to 51] | 35 [35 to 35] | 40 [35 to 51]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 1 | 1
  Male | 4 | 0 | 4
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 4 | 1 | 5
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 4 | 1 | 5
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 4 | 1 | 5

OUTCOME MEASURES:

1. Primary Outcome: Progression-free Survival Rate
Description: Progression-free survival is defined as the time from study entry to lymphoma progression or death from any cause. Proportion of patients who are progression-free and alive at 36 months will be reported. Progression is defined as appearance of any new lesions more than 1.5 cm in any axis, at least a 50% increase from nadir in sum of the product of the diameters (SPD) of any previously involved nodes or extranodal masses or the size of other lesions, or at least 50% increase in the longest diameter of any single previously identified node or extranodal mass more than 1 cm in its short axis.
Time Frame: Assessed at 36 months
Population: Only eligible and treated patients are included in this analysis
Measure: Number (95% Confidence Interval); unit: proportion of participants
Groups:
- ABVD + INRT: Induction ABVD chemotherapy: Patients receive doxorubicin hydrochloride IV, bleomycin sulfate IV, vinblastine IV over 3-5 minutes, and dacarbazine IV over 30 minutes on days 1 and 15. Treatment repeats every 28 days for 2 courses.
  PET-CT scan: Then patients undergo fludeoxyglucose F 18 (18 FDG) positron emission tomography (PET)/computed tomography (CT). If results are negative, patients receive the following treatment.
  ABVD + INRT: Patients receive doxorubicin hydrochloride, bleomycin sulfate, vinblastine, and dacarbazine as in induction chemotherapy. Treatment repeats every 28 days for 4 courses. Within 3-6 weeks after completion of chemotherapy, patients undergo involved-node radiotherapy (INRT) 5 days a week for approximately 3½ weeks.
  Doxorubicin: IV
  Bleomycin: IV
  Vinblastine: IV
  PET: fludeoxyglucose F 18 Imaging exam
  INRT: selective external radiation therapy
  Dacarbazine: IV
- ABVD + BEACOPP + INRT: Induction ABVD chemotherapy: Patients receive doxorubicin hydrochloride IV, bleomycin sulfate IV, vinblastine IV over 3-5 minutes, and dacarbazine IV over 30 minutes on days 1 and 15. Treatment repeats every 28 days for 2 courses.
  PET-CT scan: Then patients undergo fludeoxyglucose F 18 (18 FDG) positron emission tomography (PET)/computed tomography (CT). If results are positive, patients receive the following treatment.
  BEACOPP + INRT: Patients receive doxorubicin hydrochloride IV and cyclophosphamide IV over 60 minutes on day 1, etoposide IV over 60 minutes on days 1-3, procarbazine hydrochloride orally (PO) on days 1-7, prednisone PO on days 1-14, and bleomycin sulfate IV and vincristine sulfate IV on day 8. Treatment repeats every 21 days for 4 courses. Within 3-6 weeks after completion of chemotherapy, patients who achieve complete response with a negative 18FDG-PET/CT scan undergo INRT 5 days a week for approximately 3½ weeks.
  Doxorubicin: IV
  Bleomycin: IV
  Vinblastine: IV
  PET: fludeoxyglucose F 18 Imaging exam
  INRT: selective external radiation therapy
  Dacarbazine: IV
  Etoposide: IV
  Cyclophosphamide: May be given orally, IV push, or by IV infusion
  Vincristine: IV
  Procarbazine: PO
  Prednisone: PO
Arm/Group | ABVD + INRT | ABVD + BEACOPP + INRT
Number analyzed (Participants) | 4 | 1
proportion of participants | NA [NA to NA] — The study was terminated early due to slow accrual. At the time of final analysis, none of the patients were followed for 36 months so 36-month progression-free survival rate could not be reported. | NA [NA to NA] — The study was terminated early due to slow accrual. At the time of final analysis, none of the patients were followed for 36 months so 36-month progression-free survival rate could not be reported.

2. Secondary Outcome: Proportion of Patients Who Are PET Negative After Induction Treatment
Time Frame: Assessed at end of Cycle 2
Population: Only eligible and treated patients are included in this analysis
Measure: Number (90% Confidence Interval); unit: proportion of participants
Groups:
- Step 1: Induction Tx: Induction ABVD chemotherapy: Patients receive doxorubicin hydrochloride IV, bleomycin sulfate IV, vinblastine IV over 3-5 minutes, and dacarbazine IV over 30 minutes on days 1 and 15. Treatment repeats every 28 days for 2 courses.
Arm/Group | Step 1: Induction Tx
Number analyzed (Participants) | 5
proportion of participants | 0.8 [0.34 to 0.99]

3. Secondary Outcome: Progression-free Survival at 36 Months Among Patients Who Are PET Positive After Induction Treatment
Description: as for outcome 1
Time Frame: Assessed at 36 months
Population: Only patients who are PET positive are included in this analysis
Measure: Number (90% Confidence Interval); unit: proportion of participants
Arm/Group | ABVD + BEACOPP + INRT
Number analyzed (Participants) | 1
proportion of participants | NA [NA to NA] — The study was terminated early due to slow accrual. At the time of final analysis, none of the patients were followed for 36 months so 36-month progression-free survival rate could not be reported.

4. Secondary Outcome: Complete Response (CR) Rate After Induction Treatment
Description: Complete response (CR) is defined as complete disappearance of all detectable clinical evidence of disease and disease-related symptoms if present prior to therapy.
Time Frame: Assessed at end of Cycle 2
Population: Only eligible and treated patients are included in this analysis
Measure: Number (90% Confidence Interval); unit: proportion of participants
Arm/Group | Step 1: Induction Tx
Number analyzed (Participants) | 5
proportion of participants | 1.0 [0.55 to 1.0]

5. Secondary Outcome: Overall Survival
Description: Overall survival is defined as the time from study entry to death or date last known alive.
Time Frame: Assessed at 36 months
Population: Only eligible and treated patients are included in this analysis
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | ABVD + INRT | ABVD + BEACOPP + INRT
Number analyzed (Participants) | 4 | 1
months | NA [NA to NA] — Median OS was not reached. All patients were alive as of this analysis. The upper and lower limits of the 95% confidence interval were not calculable because an insufficient number of participants reached the event at the final time point for assessment. | NA [NA to NA] — Median OS was not reached. The patient was alive as of this analysis. The upper and lower limits of the 95% confidence interval were not calculable because an insufficient number of participants reached the event at the final time point for assessment.

6. Secondary Outcome: Sites of Relapse Following Combined Modality Treatment
Time Frame: Assessed at 3, 12, 18, 24 and 36 months after INRT
Population: The study was terminated early due to slow accrual. Relapse data were not collected.
Arm/Group | ABVD + INRT | ABVD + BEACOPP + INRT
Number analyzed (Participants) | 0 | 0

7. Secondary Outcome: Serum and Plasma Banking
Description: To bank serum and plasma at baseline and follow-up time point to assess the prognostic value of various markers, such as but not limited to, SCD30, IL10, CCL17, CCL22, and MDC.
Time Frame: Baseline and post cycle 2
Population: The study was terminated early due to slow accrual. Biomarker data were not collected.
Arm/Group | Step 1: Induction Tx
Number analyzed (Participants) | 0

8. Secondary Outcome: Biomarker Assessment Using Tissue Microarrays (TMAs)
Description: To create TMAs from patient tumor blocks for future biomarker assessment including but not limited to bcl-2, FOXP3, and macrophage content.
Time Frame: Baseline and relapse/progression
Population: The study was terminated early due to slow accrual. Biomarker data were not collected.
Arm/Group | Step 1: Induction Tx
Number analyzed (Participants) | 0

9. Secondary Outcome: The Association Between Thymus and Activation-related Chemokine (TARC) Levels and PET-CT Findings as Well as 3-year PFS
Description: To measure serum TARC levels pre-treatment and after two cycles of ABVD and evaluate the associations between TARC levels and PET-CT findings as well as 3-year PFS.
Time Frame: Baseline and cycle 2 for TARC assessments; 3 years for PFS
Population: The study was terminated early due to slow accrual. TARC data were not collected.
Arm/Group | Step 1: Induction Tx
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: Assessed every 4 weeks while on treatment and for 30 days after the end of treatment
Groups:
- Step 1: Induction Treatment: Induction ABVD chemotherapy: Patients receive doxorubicin hydrochloride IV, bleomycin sulfate IV, vinblastine IV over 3-5 minutes, and dacarbazine IV over 30 minutes on days 1 and 15. Treatment repeats every 28 days for 2 courses.
  PET-CT scan: Then patients undergo fludeoxyglucose F 18 (18 FDG) positron emission tomography (PET)/computed tomography (CT). Patients will be assigned to Step 2 treatments (either ABVD + INRT or BEACOPP + INRT) depending on the scan results (negative or positive).
- Step 2: ABVD + INRT: ABVD + INRT: Patients receive doxorubicin hydrochloride, bleomycin sulfate, vinblastine, and dacarbazine as in induction chemotherapy. Treatment repeats every 28 days for 4 courses. Within 3-6 weeks after completion of chemotherapy, patients undergo involved-node radiotherapy (INRT) 5 days a week for approximately 3½ weeks.
- Step 2: BEACOPP + INRT: BEACOPP + INRT: Patients receive doxorubicin hydrochloride IV and cyclophosphamide IV over 60 minutes on day 1, etoposide IV over 60 minutes on days 1-3, procarbazine hydrochloride orally (PO) on days 1-7, prednisone PO on days 1-14, and bleomycin sulfate IV and vincristine sulfate IV on day 8. Treatment repeats every 21 days for 4 courses. Within 3-6 weeks after completion of chemotherapy, patients who achieve complete response with a negative 18FDG-PET/CT scan undergo INRT 5 days a week for approximately 3½ weeks.
Arm/Group | Step 1: Induction Treatment | Step 2: ABVD + INRT | Step 2: BEACOPP + INRT
All-Cause Mortality (participants affected / at risk) | 0/6 | 0/4 | 0/1
Serious Adverse Events (participants affected / at risk) | 5/6 | 3/4 | 1/1
Other Adverse Events (participants affected / at risk) | 6/6 | 4/4 | 1/1
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Step 1: Induction Treatment (N=6) | Step 2: ABVD + INRT (N=4) | Step 2: BEACOPP + INRT (N=1)
Anemia (Blood and lymphatic system disorders) | 0 | 0 | 1
Febrile neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 1
Fatigue (General disorders) | 0 | 0 | 1
Hypothyroidism (Endocrine disorders) | 0 | 0 | 0
Infections and infestations - Other, specify (Infections and infestations) | 0 | 1 | 0
Lymphocyte count decreased (Investigations) | 1 | 1 | 0
Neutrophil count decreased (Investigations) | 4 | 3 | 1
Platelet count decreased (Investigations) | 0 | 0 | 1
White blood cell decreased (Investigations) | 0 | 1 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Step 1: Induction Treatment (N=6) | Step 2: ABVD + INRT (N=4) | Step 2: BEACOPP + INRT (N=1)
Anemia (Blood and lymphatic system disorders) | 3 | 4 | 0
Sinus tachycardia (Cardiac disorders) | 0 | 1 | 0
Chills (General disorders) | 0 | 1 | 0
Fatigue (General disorders) | 4 | 4 | 1
Fever (General disorders) | 0 | 1 | 0
Non-cardiac chest pain (General disorders) | 1 | 1 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 1 | 3 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 2 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 1 | 0
Rash acneiform (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Abdominal distension (Gastrointestinal disorders) | 1 | 1 | 0
Constipation (Gastrointestinal disorders) | 2 | 1 | 1
Dyspepsia (Gastrointestinal disorders) | 0 | 1 | 0
Dysphagia (Gastrointestinal disorders) | 1 | 0 | 0
Gastroesophageal reflux disease (Gastrointestinal disorders) | 1 | 1 | 0
Nausea (Gastrointestinal disorders) | 3 | 1 | 1
Allergic reaction (Immune system disorders) | 1 | 0 | 0
Upper respiratory infection (Infections and infestations) | 0 | 1 | 1
Carbon monoxide diffusing capacity decreased (Investigations) | 0 | 1 | 0
Creatinine increased (Investigations) | 1 | 0 | 0
Lymphocyte count decreased (Investigations) | 1 | 1 | 0
Neutrophil count decreased (Investigations) | 2 | 3 | 0
Platelet count decreased (Investigations) | 0 | 1 | 0
Weight gain (Investigations) | 1 | 1 | 0
White blood cell decreased (Investigations) | 5 | 3 | 1
Anorexia (Metabolism and nutrition disorders) | 1 | 0 | 0
Hyperglycemia (Metabolism and nutrition disorders) | 1 | 0 | 0
Hypocalcemia (Metabolism and nutrition disorders) | 0 | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Headache (Nervous system disorders) | 0 | 1 | 0
Paresthesia (Nervous system disorders) | 1 | 1 | 0
Peripheral sensory neuropathy (Nervous system disorders) | 2 | 1 | 0
Blurred vision (Eye disorders) | 1 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 | 3 | 0
Hypertension (Vascular disorders) | 1 | 0 | 0
Superficial thrombophlebitis (Vascular disorders) | 1 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less